CLINICAL TRIAL: NCT03318835
Title: An Randomized, Open-label, Phase III Study Comparing Thalidomide Combined With R-CHOP and R-CHOP in Newly Diagnosed Double-expressor Diffuse Large B-Cell Lymphoma Patients
Brief Title: Thalidomide Combined With R-CHOP in Newly Diagnosed，Untreated Double-expressor Diffuse Large B-Cell Lymphoma Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Fangfang Lv, MD, principle investigator, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDSCC LYM2017-01
Record Dates: First submitted 2017-10-11; First posted 2017-10-24 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Thalidomide
Keywords: Thalidomide; R-CHOP; diffuse large B-cell lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — R-CHOP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thalidomide combined with R-CHOP (Experimental): rituximab 375 mg/m2,ivgtt D1 cyclophosphamide 750 mg/m2 iv D2 vincristine 1.4 mg/m2 [capped at 2.0 mg], iv D2 doxorubicin 50 mg/m2 iv D2 prednisone 100 mg/m2 per day PO D2-6 Thalidomide 200mg PO QN D1-21
  Interventions: Drug: Thalidomide combined with R-CHOP
- R-CHOP (Active Comparator): rituximab 375 mg/m2,ivgtt D1 cyclophosphamide 750 mg/m2 iv D2 vincristine 1.4 mg/m2 [capped at 2.0 mg], iv D2 doxorubicin 50 mg/m2 iv D2 prednisone 100 mg/m2 per day PO D2-6
  Interventions: Drug: R-CHOP

INTERVENTIONS:
Drug: Thalidomide combined with R-CHOP — rituximab 375 mg/m2,ivgtt D1 cyclophosphamide 750 mg/m2 iv D2 vincristine 1.4 mg/m2 [capped at 2.0 mg], iv D2 doxorubicin 50 mg/m2 iv D2 prednisone 100 mg/m2 per day PO D2-6 Thalidomide 200mg PO QN D1-21
  Other Names: RT-CHOP
  Arms: Thalidomide combined with R-CHOP
Drug: R-CHOP — rituximab 375 mg/m2,ivgtt D1 cyclophosphamide 750 mg/m2 iv D2 vincristine 1.4 mg/m2 [capped at 2.0 mg], iv D2 doxorubicin 50 mg/m2 iv D2 prednisone 100 mg/m2 per day PO D2-6
  Arms: R-CHOP

SUMMARY:
The purpose of this study is to evaluate the efficacy of Thalidomide combined with R-CHOP(RT-CHOP) in newly diagnosed，untreated double-expressor Diffuse Large B-Cell Lymphoma patients (DLBCL)

DETAILED DESCRIPTION:
Double expressor lymphoma is a subtype of diffuse large B-cell lymphoma defined as having increased expression of MYC and BCL-2 and/or BCL-6 by immunohistochemistry. Patients with double-expressor lymphomas have a poor prognosis when treated with standard chemoimmunotherapy and have increased risk of progression and recurrence. The investigators conducted this study to evaluate the efficacy of Thalidomide combined with R-CHOP(RT-CHOP) in newly diagnosed double-expressed, untreated Diffuse Large B-Cell Lymphoma patients (DLBCL). Thalidomide is a kind of glutamate derivatives, which can inhibit angiogenesis by blocking bFGF and VEGF, and it can also modulate the immune system by co-stimulating T cell proliferation. In addition, thalidomide can also inhibit the IKK activity and block the activation of NF-kB. In this open-label, randomized, phase III study, we are aiming to compare Thalidomide combined with R-CHOP(RT-CHOP) and R-CHOP in newly diagnosed double-expressor Diffuse Large B-Cell Lymphoma patients (DLBCL), in order to find a potential promising way to treat this subtype of lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age range ≥18 years old
2. Eastern Cooperative Oncology Group performance status 0 to 2;
3. Newly diagnosed, untreated, histological confirmed diffuse large B cell lymphoma, non-GCB subtype, and Myc≥40% as well as Bcl-2≥70% through immunohistochemistry；
4. Measurable disease was defined as at least one lesion ≥1.5 cm in length-diameter and ≥0.5 cm in short-diameter by CT.
5. Patients have written informed consent to participate in the study.
6. Ultrasonic cardiogram showed left ventricle ejection fraction ≥ 50%, EKG showed on signs of myocardial ischemia, with no previous arrhythmia which need pharmacological intervention.
7. White blood cell ≥ 3.5×109/L, absolute neutrophil count ≥ 1.5×109/L，platelet ≥ 80×109/L，hemoglobin ≥ 90 g/L
8. total bilirubin < 1.5×upper limit of normal(ULN), ALT and AST < 1.5× ULN
9. serum creatine <1.5×ULN, and creatinine clearance rate (CCR) ≥ 30 ml/min

Exclusion Criteria:

1. Presence of CNS involvement
2. Particular kind of DLBCL，such as primary mediastinal/thymic B-cell lymphoma, elderly EBV positive DLBCL, primary cutaneous large B lymphoma.
3. History of myocardial diseases, such as congenital heart disease, pericardial disease, heart failure, myocardial infarction, coronary heart disease, valvular heart disease, myocardosis, arrhythmia.
4. History of severe chronic cutaneous diseases.
5. History of allergic asthma or severe allergic diseases.
6. Uncontrolled hypertension and diabetes.
7. History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
8. HIV, HCV, or syphilis infection；
9. Presence of active HBV infection（HBV-DNA≥104）；
10. Pregnant or lactating women
11. Previously received organ transplant
12. Having usage of Thalidomide；
13. History of deep vein thrombosis
14. Serious uncontrolled infection
15. Having contraindications to the use of large doses of hormone, such as uncontrolled hyperglycemia, gastric ulcer, mental disorder.
16. Severe neurol of mental illness, including dementia and epilepsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2017-08-22 (Actual); Primary Completion 2020-08-22 (Estimated); Study Completion 2020-08-22 (Estimated)

PRIMARY OUTCOMES:
3 year PFS | 3 years
  3 year progression free survival

SECONDARY OUTCOMES:
ORR | 6 weeks，12 weeks，18weeks
  overall response rate
OS | 3 years
  overall survival
adverse event | throughout the treatment period，up to 6 months
  adverse event related to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Fang-Fang Lv, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China